CLINICAL TRIAL: NCT01959399
Title: A Phase 1, Open-Label, Single-Sequence Drug Interaction Study to Evaluate the Effect of Multiple-Dose ASP015K on the Pharmacokinetics of Rosuvastatin in Healthy Adult Subjects
Brief Title: Drug-Drug Interaction Study Evaluating Effects of ASP015K on Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 015K-CL-PK26
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP015K
Keywords: ASP015K; healthy subjects
MeSH Terms: interventions — peficitinib; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP015K + rosuvastatin (Experimental)
  Interventions: Drug: ASP015K; Drug: Rosuvastatin

INTERVENTIONS:
Drug: ASP015K — oral tablet
Drug: Rosuvastatin — oral tablet

SUMMARY:
The purpose of this study will be to assess the effect of multiple-doses of ASP015K on the pharmacokinetics of rosuvastatin in healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Body Mass Index (BMI) range of 18.5-32.0 kg/m2, inclusive, and must weigh at least 50 kg at screening.
* Asian subject must be first generation Japanese born in Japan with both parents and four grandparents of Japanese descent and have resided outside of Japan for 5 years or less, or first generation Chinese born in China with both parents and four grandparents of Chinese descent and have resided outside of China for 5 years or less, or first generation Korean born in Korea with both parents and four grandparents of Korean descent and have resided outside of Korea for 5 years or less.
* Non-Asian subject is self-reported as White, Black or African American, and Hispanic or Latino.
* Female subject must be of non-childbearing potential (i.e., post-menopausal [defined as at least 1 year without menses] prior to screening or documented surgically sterile or status post hysterectomy [at least 1 month prior to screening]).
* Female subject must have a negative pregnancy test at screening and day -1.
* Female subject must not donate ova starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at screening and continue throughout the study period and for 90 days after final study drug administration.
* Male subject must not donate sperm from screening and throughout the study period and for 90 days after final study drug administration.
* Subject agrees not to participate in another investigational study while on treatment.
* Subject must be capable of swallowing multiple tablets.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months before screening assessment or breast feeding within 3 months before screening.
* Subject has a known or suspected hypersensitivity to rosuvastatin, ASP015K, or any components of the formulations used.
* Subject has had a previous intolerance or adverse reaction to a statin therapy.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has any history or evidence of any clinically significant cardiovascular, gastro intestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy, as judged by the Investigator or designee.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to day -1.
* Subject has a mean pulse < 40 or > 90 beats per minute (bpm); mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (measurements taken in triplicate after subject has been resting in sitting position for at least 5 minutes at screening and day -1.
* Subject has used any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g. St. John's Wort) in the 2 weeks prior to study drug administration, with the exception of hormone replacement therapy (HRT) and intermittent acetaminophen (to a maximum of 2 g/day).
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine containing products in the past 6 months prior to screening.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits).
* Subject has a positive test for alcohol, drugs of abuse, or cotinine at screening or day -1.
* Subject has used any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to day -1.
* Subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic check-in on day -1.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg) (total), anti hepatitis A virus (Ig M), anti-hepatitis C virus, anti-hepatitis B core, or anti HIV type 1 or type 2 at screening.
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives of the drug, whichever is longer, prior to screening.
* Subject has a positive tuberculosis (TB) skin test, Quantiferon Gold test or T-SPOT® test at screening.
* Subject has received any vaccine within 60 days prior to study drug administration.
* Subject has had major gastrointestinal surgery or has a medical condition which may inhibit the absorption and/or metabolism of study drug.
* Subject anticipates an inability to abstain from xanthine (e.g., caffeine), grapefruit, Seville blood oranges (including marmalade), star fruit, or any products containing these items from 72 hours prior to day -1 and throughout the duration of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameter for rosuvastatin: AUClast | Days 1 and 10
  Area under the curve to the last measurable time
Pharmacokinetic parameter for rosuvastatin: AUCinf | Days 1 and 10
  Area under the curve to the infinity
Pharmacokinetic parameter for rosuvastatin: Cmax | Days 1 and 10
  Maximum Concentration

SECONDARY OUTCOMES:
Composite of pharmacokinetic parameters for rosuvastatin: time after dosing when Cmax occurs (tmax), apparent-terminal elimination half-life (t1/2), apparent volume of distribution (Vz/F), apparent plasma clearance (CL/F) | Days 1 and 10
Composite of PK parameters for ASP015K: Area under the curve in the dosing interval (AUCtau), Maximum Concentration (Cmax), time after dosing when Cmax occurs (tmax), apparent volume of distribution (Vz/F), apparent plasma clearance at steady (CLss/F) | Days 9 and 10
Pharmacokinetic parameter for ASP015K: Ctrough | Days 7-10
  Plasma concentration immediately before the next administration of study drug
Pharmacokinetic parameter for ASP015K metabolites: Ctrough | Days 7-10
  Plasma concentration immediately before the next administration of study drug
Composite of pharmacokinetic parameters for ASP015K metabolites: Area under the curve in the dosing interval (AUCtau), Maximum Concentration (Cmax), time after dosing when Cmax occurs (tmax) | Days 9 and 10
Safety assessed adverse events, clinical laboratory evaluations, 12-lead ECG measurements, physical examination and vital sign measurements | Day 1-14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- PAREXEL - Early Phase Unit, Glendale, California, United States

REFERENCES:
- [Derived] Zhu T, Parker B, Wojtkowski T, Nishimura T, Garg JP, Han D, Fisniku O, Keirns J. Drug Interactions Between Peficitinib, an Orally Administered, Once-Daily Janus Kinase Inhibitor, and Rosuvastatin in Healthy Subjects. Clin Pharmacokinet. 2017 Jul;56(7):747-757. doi: 10.1007/s40262-016-0474-4. PMID 27878567